CLINICAL TRIAL: NCT06883253
Title: Establishing Individualized Step Cadence Thresholds for Moderate-to-Vigorous Intensity in Taiwanese Obese Young Adults: A Cross-Sectional Study
Brief Title: Individualized Cadence Thresholds for Moderate-to-Vigorous Intensity in Obese Taiwanese Young Adults
Status: Completed | Type: Observational
Sponsor: Chinese Culture University (Other)
Responsible Party: Principal Investigator, TSUNG-LIN CHIANG, Researcher, National Science and Technology Council, Taiwan
Other Study IDs: No. 105-2815-C-034-028-H; 105-2815-C-034-028-H (Other Grant/Funding Number: National Science and Technology Council, Taiwan)
Record Dates: First submitted 2025-03-06; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Body Composition; Cadence; Physical Activity Intensity
Keywords: Obese; Oxygen consumption; Metabolic equivalent; Steps per minute; Step rete thresholds
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Obese Young Adults: This study includes 48 obese young adults, approximately 20 years old, with 28 males and 20 females.
  Interventions: Behavioral: treadmill walking

INTERVENTIONS:
Behavioral: treadmill walking — all participants walking at increasing speeds on a treadmill

SUMMARY:
This study aims to determine the step cadence thresholds for moderate-to-vigorous physical activity (MVPA) in obese young adults. It examines the relationship between body composition and step cadence required to achieve moderate-intensity physical activity (MPA, 3 METs), MPAyoung (4.8 METs), and vigorous physical activity (VPA, 6 METs).

DETAILED DESCRIPTION:
Background: This study examined the relationship between body composition and Moderate-to-Vigorous Physical Activity (MVPA) cadence in obese individuals and establish cadence thresholds for moderate-intensity physical activity (MPA) (3 metabolic equivalents [METs]), MPAyoung (4.8 METs), and vigorous physical activity (VPA) (6 METs).

Methods: This study recruited 48 obese young adults who did not regularly engage in exercise. Exclusion criteria included a history of smoking, hypertension, diabetes, cardiovascular or respiratory diseases, neuromuscular or musculoskeletal disorders, or any condition deemed unsuitable for exercise by a physician. The study protocol was approved by the Fu Jen University Institutional Review Board for Human Research (Approval Number: C105137). All participants were fully informed about the study procedures and provided written informed consent prior to participation.

Anthropometrics and Body Composition Measurements Participants arrived at the lab fasted for a minimum of 3 hours, abstained from exercise for 12 hours, avoided caffeine for 6 hours, and refrained from alcohol consumption for 12 hours. Data collection for each subject occurred during the morning hours, as close as possible to awakening from sleep (i.e., from 7:00 AM to 10:00 AM). Height was measured using a digital stadiometer accuracy nearest to ± 0.1 cm (Kongho-Super View, Kong Ho Instruments Co., Ltd., New Taipei, Taiwan). Body composition was assessed using bioelectrical impedance analysis (BIA) with the InBody 720 device (Biospace Co., Ltd., Seoul, South Korea). Skin resistance was measured through an eight-point tactile-electrode system at different frequencies (1 kHz, 5 kHz, 50 kHz, 250 kHz, 500 kHz, 1 MHz). Lean body mass and fat mass were determined from the impedance values using the manufacturer's regression equations, based on the principle that different tissues have varying water content and, consequently, different electrical conductivity 30. The components used in further analysis included weight, body mass index (BMI), body fat mass (BFM), body fat percentage (FAT), visceral fat area (VFA), and skeletal muscle mass (SMM).

Incremental Submaximal Exercise Testing Protocol Participants were instructed to refrain from vigorous exercise, smoking, and the consumption of caffeine-containing foods and beverages for 24 hours prior to the experiment. During the test, each participant was equipped with a gas analyzer (MetaMax 3B, Cortex, Leipzig, Germany) and a heart rate monitor (Polar H10, Electro Oy, Kempele, Finland). The protocol began with a 10-minute seated rest period to measure resting oxygen consumption. Subsequently, participants completed an incremental submaximal treadmill walking test consisting of five stages, with speeds set at 3.2, 4.0, 4.8, 5.6, and 6.4 km/h. Each stage lasted 5 minutes, and participants were instructed to maintain a natural walking pattern throughout the test. Oxygen consumption was continuously recorded during the exercise phases using the gas analyzer, while the total step count for each stage was captured using a video camera.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19-21 years
* BMI classified as obese (≥27 kg/m²)
* Able to walk on a treadmill without assistance

Exclusion Criteria:

* Presence of metabolic, cardiovascular, or musculoskeletal disorders
* History of bariatric surgery
* Current participation in structured exercise program

Ages: 19 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of obese young adults aged approximately 20 years. Participants include both males and females, with a BMI classified as obese (≥27 kg/m²). The study aims to examine the relationship between step cadence and metabolic equivalents during walking.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
Step Cadence Thresholds for Moderate-to-Vigorous Physical Activity in Obese Young Adults | Day 1
  This study examines the step cadence thresholds required to achieve moderate-to-vigorous physical activity (MVPA) in obese young adults. The primary outcome measure is the step cadence corresponding to 3 METs (MPA), 4.8 METs (MPAyoung), and 6 METs (VPA), determined through indirect calorimetry during incremental treadmill walking.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Culture University, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiang TL, Lin YC, Chen C, Chan SH, Ye YY, Hsu CH, Su PW, Wu HJ. Individualized walking cadence thresholds of moderate to vigorous intensity for Taiwanese obese young adults. BMC Public Health. 2025 Oct 14;25(1):3471. doi: 10.1186/s12889-025-24805-7. PMID 41088002